CLINICAL TRIAL: NCT01592643
Title: Post Photorefractive Keratectomy (PRK) Use of an Eye Shield for Maintaining Vision and Mitigating Pain
Acronym: Nexis-CS0032
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22760
Record Dates: First submitted 2012-04-19; First posted 2012-05-07 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Pain; Vision Nearsighted
Keywords: Corneal shield; PRK; Myopia; Pain; Vision
MeSH Terms: conditions — Pain; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eye shield (Experimental): Participants receive eye shield during PRK surgery
  Interventions: Device: Eye Shield

INTERVENTIONS:
Device: Eye Shield — The thin shield is made of silicone. The materials used to make the corneal shield all have a history of use in medical devices, contact lenses, and/or corneal shields and have been used safely in the eye.
  Other Names: Nexis Vision corneal shield

SUMMARY:
The purpose of this research is to determine if an investigational thin shield over the cornea can safely and effectively reduce or eliminate pain following Post Photorefractive Keratectomy (PRK).

The thin shield is made of silicone. The materials used to make the corneal shield all have a history of use in medical devices, contact lenses, and/or corneal shields and have been used safely in the eye.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion criteria.

* Subjects age 18 and older with healthy eyes.
* Nearsightedness between -0.50 diopters and -11.00 diopters with or without astigmatism of up to 3.50 diopters.

Exclusion criteria.

* Subjects under the age of 18.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectactic eye disorders.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.
* Any other anterior segment abnormality other than that associated with PRK
* Any abnormalities associated with the eye lids
* Uncontrolled blepharitis or dry eye
* Prior laser treatment of the retina
* Any ophthalmic surgery performed within three (3) months prior to study excluding PRK or LASIK
* Diagnosis of glaucoma
* Active diabetic retinopathy
* Clinically significant inflammation or infection within six (6) months prior to study
* Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator
* Participation in any study involving an investigational drug within the past 30 calendar days, or ongoing participation in a study with an investigational material
* Intolerance or hypersensitivity to topical anesthetics, antibiotics, steroids or any other pharmaceuticals that may be used pre and post surgically Specifically known intolerance or hypersensitivity to contact lenses or any component of the investigative material
* A medical condition, serious concurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up
* Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

REFERENCES:
- [Result] Sales CS, Manche EE. Prospective evaluation of a novel silicone corneal shield after PRK: 6-month efficacy, safety, and predictability outcomes. Clin Ophthalmol. 2019 Jan 7;13:115-121. doi: 10.2147/OPTH.S183120. eCollection 2019. PMID 30662255

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Eye Shield
Started | 30; 45 Eyes
Completed | 30; 45 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Eye Shield
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pain Score of Four or Greater. Score Range: 0-10, Higher Score Corresponds to More Pain.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Eye Shield
Number analyzed (Participants) | 30
Participants | 0

2. Secondary Outcome: Mean Change in Uncorrected Visual Acuity
Description: LogMAR uncorrected visual acuity. Values closer to zero indicate improved vision
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Eye Shield
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 45
logMAR
  Baseline | 1.34 (0.55)
  Month six | -0.06 (0.11)

ADVERSE EVENTS:
Time Frame: Six months
Arm/Group | Eye Shield
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT01592643/Prot_SAP_000.pdf